CLINICAL TRIAL: NCT06545071
Title: Autonomous Digital CBT Intervention for Opioid Use Disorder in Individuals With Co-Occurring Internalizing Disorders - UG3
Brief Title: Autonomous Digital CBT Intervention for Opioid Use Disorder in Individuals With Co-Occurring Internalizing Disorders
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 32774; UG3DA059414 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder; Anxiety; Depression
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Behavioral: NEAT-O program

INTERVENTIONS:
Behavioral: NEAT-O program — NEAT-O's curriculum is designed to interrupt the cycle of negative emotions and opioid use through a multifaceted approach encompassing physiological, psychological, and behavioral strategies. The program includes interactive modules that capture the core therapeutic components of CBT and teach skills to support OUD recovery.

SUMMARY:
The primary objective of this protocol is to implement the UG3 phase (Phase 1) of a National Institute on Drug Abuse (NIDA) UG3/UH3 grant (RFA-DA-23-049). This phase is dedicated to the pilot testing of NEAT-O, a digital Cognitive Behavioral Therapy (CBT) program tailored for individuals with opioid use disorder (OUD) and concurrent anxiety or mood disorders - collectively referred to as internalizing disorders (INTDs). NEAT-O is based on an empirically supported CBT framework, specifically modified to address the complexities of comorbidity in substance use disorders (SUDs). This pilot study will evaluate the usability and acceptability of NEAT-O in 15 participants with OUD, with the goal of refining the program's content and delivery methods. The results of the pilot study will inform a comprehensive RCT in the UH3 Phase (Phase 2) (N=300). Progression to the UH3 phase, with its funding, depends on meeting milestones in Phase 1 including demonstrating protocol adherence and the program's acceptability and usability.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 to 65
* Current DSM-5 diagnosis of OUD (confirmed during MINI 7 interview)
* Current DSM-5 diagnosis of panic disorder with or without agoraphobia (PD/Ag) generalized anxiety disorder, social anxiety disorder, or major depression (confirmed during MINI 7 interview)
* Currently in treatment for OUD using MOUD
* Access to an internet-enabled smartphone for the duration of the study
* Currently residing in the United States
* Provision of informed consent

Exclusion Criteria:

* Current diagnosis of psychosis
* Current institutionalization (e.g., jail, hospital)
* Self-reported pregnancy
* Non-English Speakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 45 days
  Measured by the completion rate of NEAT-O modules, app usage frequency, modules accessed, and session length (after each module). Interaction frequency and module completion rates will be quantified using frequency counts and percentages.
Usability | 45 days
  Evaluated using the System Usability Scale (SUS) to assess effectiveness, efficiency, and satisfaction. The SUS is a well-validated questionnaire with 10 items. 27 Scores of 70 or above on the SUS are considered acceptable (Post-Tx).
Attractiveness and Information Quality | 45 days
  The Mobile Application Rating Scale (MARS) will be used to evaluate the attractiveness and information quality of NEAT-O. Scores of 3 or higher (out of a maximum score of 5) on the MARS are generally considered acceptable and indicate that the app has a high level of overall quality and content (after each module).

SECONDARY OUTCOMES:
Feasibility of EMA Collection Among Individuals with OUD | 45 days
  Compliance with the EMA procedure will be assessed by tracking the number of days EMA prompts are completed as well as the average number of prompts completed per day using frequency counts and percentages.
Recruitment and Retention Metrics | 45 days
  Recruitment effectiveness and participant retention will be monitored through descriptive statistics, including counts, percentages, and adherence rates to the recruitment timeline.
Preliminary Efficacy Indicators | 45 days
  Patterns of opioid use (e.g., EMA data, Pre and Post-Tx measures), quality of life (WHODAS 2.0 scores), measures derived from the neurobiological domains of the addiction. These measures will be analyzed using descriptive and inferential statistics to identify early patterns and improvements.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States